CLINICAL TRIAL: NCT07321470
Title: A Single Center Prospective Randomized Trial of Complete vs. Postoperative Nasogastric Tube Omission in Pancreaticoduodenectomied Patients
Brief Title: Complete vs. Postoperative Nasogastric Tube Omission in Pancreaticoduodenectomied Patients
Acronym: PDNONG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202510174RINB
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Peri-ampullary Tumor
Keywords: Pancreaticoduoidenctomy, Nasogastric tube

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONGT (Experimental): Intraoperative decompression of distended stomach by thick needle suction
  Interventions: Other: Thick needle suction
- PONGT (Active Comparator): Intraoperative decompression of distended stomach through preoperatively-placed NG tube
  Interventions: Other: PONGT

INTERVENTIONS:
Other: Thick needle suction — Intraoperative decompression of distended stomach by thick needle suction
  Arms: CONGT
Other: PONGT — Decompression of distended stomach through preoperatively-placed NG tube
  Arms: PONGT

SUMMARY:
Enhanced recovery after surgery (ERAS) programs recommend early removal of a nasogastric tube ( NGT) after operation has been suggested in elective major abdominal surgery, such as colorectal3, gastric4, and hepatic surgery5. However, in spite of immediate removal after operation, NGT is still worldwide routinely inserted before major abdominal surgery. The rationale to insert NGT before operation include prevention of aspiration pneumonia during anesthesia and use for decompression of the distended stomach induced by mask bagging during anesthesia induction. However, the risk of aspiration pneumonia during intubation is so low that even American Society of Anesthesiology (ASA) guidelines for preoperative fasting guideline suggest continuing a clear carbohydrate supplement drink up to 2 hours prior to operation for decreasing the fasting period.6 Indeed, musk bagging during anesthesia occasionally will distend the stomach with air to a great extent to make the operation difficult. Besides, for anatomic reasons, the insertion of NGTs into anesthetized and intubated patients during operation for decompression of distended stomach can be very challenging.7 Therefore, in spite, distended stomach occur only occasionally and insertion of a NGT into conscious patients cause a lot of discomfort, most centers adopt policy to insert it before operation. But, it is not necessary to insert a NGT during operation for decompression of distended stomach. Instead, investigators developed a novelty method to decompress distended stomach intraoperatively by thick needler suction. With this new technique, 578 PDs have been successfully performed with complete omission of NGT (CONGT)8 and none of them needed the intraoperative insertion of NGT for decompression of encountered distended stomach. Based on the excellent results of previous study, investigators further propose a prospective randomized trial to compare complete versus postoperative omission of nasogastric tube in pancreaticoduodenectomied patients.

The complete omission of NGT (CONGT) study will be a prospective, single-center randomized controlled trial with 2 groups comparing rate of postoperative complications between pancreaticoduodenectomied patients with complete (CONGT) or traditional postoperative omission of NGT (PONGTR). Key inclusion criteria will be patients between 20 and 75 years of age requiring PD for benign or malignant disease of the biliopancreatic confluence and without symptoms or signs of intestinal obstruction (such as vomiting, presence of nasogastric tube). The primary end point will be the occurrence of a Clavien-Dindo classification grade II or higher postoperative complication. The secondary outcomes will be occurrence of pulmonary complications; occurrence of delayed gastric emptying; occurrence of pancreatic fistula; occurrence of biliary fistula or hemorrhage; the need for surgical reintervention; NGT reinsertion rate; 90-day mortality rate; length of hospital stay; and the readmission rate until 90 days after surgery.

216 patients will be required to have 80 per cent power to test the non-inferiority of CONGT compared with PONGT, with a non-inferiority margin of 20 per cent. Assuming a 10 per cent dropout rate, the final planned sample size will be 240 patients. Analyses will be conducted with the intent-to-treat population.

As the most destructive abdominal surgery, PD should be the last type of abdominal surgical procedure performed with CONGT because of associated highest rate of delayed gastric emptying. Therefore, positive results of this study could be implied to millions of patients undergoing abdominal surgery and avoid their NGT-insertion-associated discomfort.

DETAILED DESCRIPTION:
Routine use of nasogastric tubes (NGT) during abdominal surgery, historically intended to hasten bowel function return, prevent pulmonary complications, and reduce risks like anastomotic leakage, has been found largely ineffective.1 Early removal or selective use of NGT (postoperative omission of NGT, [PONGT]) is considered safer and leads to better outcomes including shorter hospital stay and less pulmonary complications.2 Therefore Enhanced recovery after surgery (ERAS) programs recommend early removal of an NGT has been suggested after major abdominal surgery, such as colorectal3, gastric4, and hepatic surgery5. However, in spite of immediate removal after surgery, NGT is still worldwide routinely inserted before abdominal surgery. The rationales to use preoperative NGT include 1. prevention of aspiration pneumonia during anesthesia and 2. use for decompression of the distended stomach induced by mask bagging during anesthesia induction. However, the risk of aspiration during anesthesia is so low that American Society of Anesthesiology (ASA) guidelines for preoperative fasting even suggest continuing a clear carbohydrate supplement drink up to 2 hours prior to operation for decreasing the fasting period.6 Musk bagging during anesthesia occasionally will distend the stomach with air to a great extent to make the operation difficult. Besides, for anatomic reasons, the insertion of NGTs into anesthetized and in tubated patients during operation for decompression of distended stomach can be very challenging.7 Therefore, most centers adopt policy to insert the NGT before operation. However, insertion of a NGT before operation into patients with clear consciousness causes a lot of discomfort. But, as shown in investigators' previous report8, instead of NGT, the distended stomach encountered during operation could be alternately decompressed through thick needle suction. In that case, the preoperative insertion of NGT could also be avoided. Therefore, the NGT could be omitted throughout the whole perioperative course of abdominal surgery, i.e. complete omission of NGT (CONGT).

Pancreaticoduodenectomy (PD) is the most destructive abdominal surgery with highest rate of postoperative complications. 9-11 Notably, among the common PD-related complications, delayed gastric emptying (DGE) remains the most common complication associated with the need for NGT placement, and its prevalence rate ranges from 3.2% to 59.0%. 12, 13 Nevertheless, more and more centers14-18 also adopt policy of removal of NGT immediate after PD (PONGT). But again, NGT is still widely used before and during PD. Theoretically, PD should be the last type of abdominal surgical procedure performed with complete omission of NGT because of associated highest rate of delayed gastric emptying. However, as shown ininvestigators' recent report, 578 PDs have been safely performed with complete omission of NGT.8 None of them needed the intraoperative insertion of NGT to decompress distended stomach. Moreover, there was significant less pulmonary complication in patients operated with CONGT compared to those operated with NGT omission only after operation. Based on the excellent results of previous study, investigators further propose a single center prospective randomized trial to compare complete versus postoperative omission of nasogastric tube in pancreaticoduodenectomied patients.

Study Design and Participants： The complete omission of NGT (CONGT) study will be a prospective, single-center RCT with 2 groups (PD performed with CONGT or PONGT) comparing rate of occurrence of postoperative complications (trial protocol in Supplement 1). The study will be performed in accordance with good clinical practice guidelines and the principles of the Declaration of Helsinki.19 This study will follow the Consolidated Standards of Reporting Trials (CONSORT) reporting guideline. The study protocol will be approved by Ethics Committee of National Taiwan University Hospital. Written informed consent will be obtained from all patients in accordance with the Declaration of Helsinki. No one will receive compensation or be offered any incentive for participating in this study. All patients scheduled for PD at the National Taiwan University Hospital will be screened and assessed for CONGT trial eligibility. Key inclusion criteria will be patients between 20 and 75 years of age requiring PD for benign or malignant disease of the biliopancreatic confluence and without symptoms or signs of intestinal obstruction (such as vomiting, presence of nasogastric tube). Key exclusion criteria will be previous gastric or esophageal surgery, severe comorbidities, such as end-stage kidney disease (creatinine clearance, <15 mL/min/1.73m2; to convert to mL/s/m2, multiply by 0.0167), documented chronic respiratory disease, heart failure (New York Heart Association class III or higher), pregnancy, nursing mothers, and persons under legal protection (guardianship).

Surgery All PD procedures will be performed by senior pancreatic surgeons (YWT, CHW) via laparotomy. A standard lymph node dissection will be performed, including the right lateral and superior aspect of the mesenteric superior artery and a paraaortic lymph node picking under the left renal vein in case of pancreatic head carcinoma. All reconstruction procedures will be standardized with pancreatojejunostomy and antecolic gastrojejunal or duodenojejunal anastomosis. Pancreatojejunostomy will be performed by an end-to-side one-layer pancreaticojejunostomy with a trans-anastomotic internal stent in the pancreatic duct using a suitable pediatric feeding tube as previously described.20 Vascular (vein or artery) resection will be performed when necessary. Three 7-mm Jackson-Pratt® drains will routinely be placed after all anastomoses [pancre- aticojejunal (PJ) reconstruction, hepaticojejunostomy (HJ) reconstruction, and antecolic gastro- /duodenojejunal reconstruction in sequential order)]. One will be placed near the PJ, another near the HJ, and the other at the left retroperitoneal cavity to precisely define the postoperative pancreatic fistula according to the International Study Group of Pancreatic Fistula (ISGPF) classification.21 Anesthesia will be administered according to the routine institution protocol used at the National Taiwan University Hospital. General anesthesia will be induced with administration of intravenous (IV) propofol, sufentanil citrate, and cisatracurium and maintained with either sevoflurane or desflurane. Continuous IV ketamine hydrochloride will be administered intraoperatively at antihyperalgesic doses. Self-paid epidural with ropivacaine hydrochloride for 24 to 48 hours will be given at patients' choice. Postoperative nausea and vomiting prevention was ensured with administration of IV dexamethasone sodium phosphate, 8 mg, during induction of anesthesia and then with IV droperidol or IV ondansetron hydrochloride according to the Apfel score.22 For antibiotic prophylaxis, IV cefmetazole sodium, 2 g, will be administered during induction of anesthesia and followed by administration of 1 g IV every 3 hours during surgery.

Management of NGT Included patients will be randomized into CONGT and PONGT groups in 1 : 1 ratio. Patients in the PONGT group will have a 14- French NGT inserted before the operation and removed at completion of operation at operating room. In contrast, for patients in CONGT group, no NGT tube will be inserted before or during operation. Distended stomach encountered during operation will be decompressed by preoperatively-placed NGT in PONGT and by thick needle suction in CONGT group patients. Patients in both groups will be allowed to drink 300-500 mL of liquids on postoperative day 1, and afterwards a soft diet will be given for 2 days. If this well tolerated, increasing amounts of solid food will be given. The NGT will be reinserted if the patient later vomits a volume of more than 300 mL or more than one occasion. Reinserted tubes will be removed if the reflux is less than 200 mL per 24 h, and oral feeding (initially with a liquid diet) will be tried again.

Postoperative Care Postoperative analgesia will be multimodal and include administration of paracetamol, celebrex, or epidural analgesia with ropivacaine for 24 to 48 hours and morphine patient-controlled analgesia as rescue analgesia. Mobilization will be begun as soon as possible (usually the next day after operation). Drainage tubes will be removed in the absence of hemorrhage or postoperative pancreatic fistula on day 4 or 5 after surgery, depending on the amylase level.

Outcomes Members of the surgical staff, not involved in the trial, will record postoperative complications. The postoperative course of each patient will be closely monitored. The day of passage of flatus and oral food intake, and length of hospital stay will be recorded. Mortality, abdominal complications, pulmonary complications (pneumonia, atelectasis), postoperative fever, nausea, and vomiting, tube reinsertion, discomfort from the tube (ear pain, nasal soreness, painful swallowing), and duration of reinserted NGT will be noted. According to the recommendation by the International Study Group of Pancreatic Surgery (ISGPS)12, gastroparesis will be defined as the need for the need to reinsert the NGT for persistent vomiting after surgery. The severity of gastroparesis will be classified by the ISGPS definition12 as grade A: NGT required for 4-7 days or reinsertion after postoperative day (POD) 3 or inability to tolerate solid oral intake by POD 7; grade B: NGT required for 8-14 days or inability to tolerate solid oral intake by POD 14; grade C: NGT required for >14 days or inability to tolerate solid food by POD 21. Again, according to the International Study Group definition, postoperative pancreatic fistula will be defined as output via an operatively placed drain (or a subsequently placed percutaneous drain) of any measurable volume of drain fluid on or after POD 3, with an amylase content greater than three times the upper normal serum value.21 Postoperative bleeding will also be graded using ISGPS definitions.23 All infectious complications will be proven by microbiological analysis and positive fluid The primary end point will be the occurrence of a Clavien-Dindo classification grade II or higher postoperative complication (range I to V, with higher scores indicating more severe complication).24 The secondary outcomes will be occurrence of pulmonary complications (including atelectasis, pleural effusion, and pneumonitis); occurrence of delayed gastric emptying (based on the International Study Group on Pancreatic Surgery guidelines as A, B, or C, with increasing clinical severity12); occurrence of pancreatic fistula (classified according to the ISGPF classification as A, B, or C, with increasing clinical severity21); occurrence of biliary fistula or hemorrhage; the need for surgical reintervention; NGT reinsertion rate (time and causes); 90-day mortality rate; length of hospital stay; and the readmission rate until 90 days after surgery. Patients will be followed up until 90 days after surgery (on days 30 and 90) using standardized case report forms completed by local study coordinators and then verified by an independent clinical research associate as stated in the protocol. Preoperative data will be collected by the investigator or by an independent clinical research associate as stated in the protocol (trial protocol in Supplement 1). Data will be collected from case report forms and entered an electronic database, with data accuracy double checked. Medical records and case report forms will be reviewed to resolve missing or implausible data.

Reinsertion of NGT and Safety Patient safety will be monitored by a board that could stop the study if adverse events occurred or more than 8 of the first 10 patients required NGT replacement. To avoid bias, surgery will be performed only by 2 senior surgeons (Y.W.T., C.H.W.) with substantial experience in pancreatic resection, including PD.

Statistical Analysis

Sample size estimation:

Given a one-sided α level of 2.5 per cent and assuming a rate of 54 per cent for complication of Clavien-Dindo classification grade II or higher, based on authors' pilot data,17 216 patients will be required to have 80 per cent power to test the non-inferiority of CONGT compared with PONGT, with a non-inferiority margin of 20 per cent. This non-inferiority margin is based on a previous study15 and the pilot data, which showed that the rate of complications of Clavien-Dindo classification grade II or higher with complete and postoperative omission of NGT in pancreaticoduodenectomied patients were approximately 38.2 and 53.8 per cent respectively. The non-inferiority margin will be set at 20 per cent to avoid loss of more than half of the benefit of PONGT over CONGT. Assuming a 10 per cent dropout rate, the final planned sample size will be 240 patients. Analyses will be conducted with the intent-to-treat population (Figure 1 Flowchart). A randomization list will be produced randomly with a block size of two.

The primary end point will be compared between the 2 groups with the χ2 test. Secondary end points will be compared with t tests or Mann-Whitney tests as appropriate for continuous variables, and with χ2 tests or Fisher exact tests as appropriate for qualitative variables. For primary and secondary outcomes, risk ratios with 95% Cis will be calculated for qualitative variables. Qualitative variables will be expressed as number of observations (percentages), and continuous variables will be expressed as mean (SD) values or as median values with interquartile ranges (IQRs). Patients who do not reach experiment end points (such as those with unplanned readmission or diet tolerance), owing to early postoperative death, will be excluded from the analysis (detailed in the respective tables). Investigators will also conduct an exploratory analysis to identify risk factors for NGT reinsertion in the CONG group to identify risk factors that could help better identify patients who would or would not need an NGT before and during surgery. All analyses were 2-sided, and the threshold for statistical significance will be set at P < .05. Analyses will be performed with R statistical software, version 3.6.3 (The R Project for Statistical Computing).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of benign or malignant disease of the biliopancreatic confluence.
* Age between 20 and 75 years of age

Exclusion Criteria:

* previous gastric or esophageal surgery
* end-stage kidney disease (creatinine clearance, <15 mL/min/1.73m2; to convert to mL/s/m2, multiply by 0.0167)
* documented chronic respiratory disease
* heart failure (New York Heart Association class III or higher)
* pregnancy
* nursing mothers
* persons under legal protection (guardianship).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
occurrence of a Clavien-Dindo classification grade II or higher postoperative complication | within 90 days after operation

SECONDARY OUTCOMES:
pulmonary complications | within 90 days after operation
  atelectasis, pleural effusion, and pneumonitis
delayed gastric emptying | Within 90 days after operation
  The inability to return to a standard diet by the end of the first postoperative week and includes prolonged nasogastric tube intubation of the patients. Based on the International Study Group on Pancreatic Surgery guidelines, delayed gastric emptying will be graded as A, B, or C, with increasing clinical severity
pancreatic fistula | within 90 days after operation
  A drain output of any measurable volume of fluid with amylase level > 3 times the upper limit of institutional nornal serum amylase activity. Based onto the ISGPF classification, pancreatic fistula will be further graded as A, B, or C, with increasing clinical severity
biliary fistula | within 90 days after operation
  Biliary fistula: a drain output of any measurable volume of fluid with an bilirubin level > 3 times the upper limit of institutional normal serum bilirubin activity.
the need for surgical reintervention | within 90 days after operation
NGT reinsertion rate | within 90 days after operation
length of hospital stay | within 90 days after operation
  Length of hospital stay after operation with all drainage tubes removed

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Result] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Result] Wu JM, Lin YJ, Wu CH, Kuo TC, Tien YW. Novel Non-duct-to-Mucosa Pancreaticojejunostomy Reconstruction After Pancreaticoduodenectomy: Focus on the Occurrence of Post-pancreatectomy Hemorrhage and Intra-abdominal Abscess. Ann Surg Oncol. 2023 Aug;30(8):5063-5070. doi: 10.1245/s10434-023-13114-1. Epub 2023 Feb 18. PMID 36808588
- [Result] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Result] Bergeat D, Merdrignac A, Robin F, Gaignard E, Rayar M, Meunier B, Beloeil H, Boudjema K, Laviolle B, Sulpice L. Nasogastric Decompression vs No Decompression After Pancreaticoduodenectomy: The Randomized Clinical IPOD Trial. JAMA Surg. 2020 Sep 1;155(9):e202291. doi: 10.1001/jamasurg.2020.2291. Epub 2020 Sep 16. PMID 32667635
- [Result] Park JS, Kim JY, Kim JK, Yoon DS. Should Gastric Decompression be a Routine Procedure in Patients Who Undergo Pylorus-Preserving Pancreatoduodenectomy? World J Surg. 2016 Nov;40(11):2766-2770. doi: 10.1007/s00268-016-3604-0. PMID 27272269
- [Result] Kleive D, Sahakyan MA, Labori KJ, Lassen K. Nasogastric Tube on Demand is Rarely Necessary After Pancreatoduodenectomy Within an Enhanced Recovery Pathway. World J Surg. 2019 Oct;43(10):2616-2622. doi: 10.1007/s00268-019-05045-4. PMID 31161355
- [Result] Flick KF, Soufi M, Yip-Schneider MT, Simpson RE, Colgate CL, Nguyen TK, Ceppa EP, House MG, Zyromski NJ, Nakeeb A, Schmidt CM. Routine Gastric Decompression after Pancreatoduodenectomy: Treating the Surgeon? J Gastrointest Surg. 2021 Nov;25(11):2902-2907. doi: 10.1007/s11605-021-04971-w. Epub 2021 Mar 26. PMID 33772404
- [Result] Kunstman JW, Klemen ND, Fonseca AL, Araya DL, Salem RR. Nasogastric drainage may be unnecessary after pancreaticoduodenectomy: a comparison of routine vs selective decompression. J Am Coll Surg. 2013 Sep;217(3):481-8. doi: 10.1016/j.jamcollsurg.2013.04.031. Epub 2013 Jul 25. PMID 23891073
- [Result] Panwar R, Pal S. The International Study Group of Pancreatic Surgery definition of delayed gastric emptying and the effects of various surgical modifications on the occurrence of delayed gastric emptying after pancreatoduodenectomy. Hepatobiliary Pancreat Dis Int. 2017 Aug 15;16(4):353-363. doi: 10.1016/S1499-3872(17)60037-7. PMID 28823364
- [Result] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Result] Wu JM, Ho TW, Yen HH, Wu CH, Kuo TC, Yang CY, Tien YW. Endoscopic Retrograde Biliary Drainage Causes Intra-Abdominal Abscess in Pancreaticoduodenectomy Patients: An Important But Neglected Risk Factor. Ann Surg Oncol. 2019 Apr;26(4):1086-1092. doi: 10.1245/s10434-019-07189-y. Epub 2019 Jan 23. PMID 30675700
- [Result] Akashi M, Nagakawa Y, Hosokawa Y, Takishita C, Osakabe H, Nishino H, Katsumata K, Akagi Y, Itoi T, Tsuchida A. Preoperative cholangitis is associated with increased surgical site infection following pancreaticoduodenectomy. J Hepatobiliary Pancreat Sci. 2020 Sep;27(9):640-647. doi: 10.1002/jhbp.783. Epub 2020 Jul 2. PMID 32506646
- [Result] Costi R, De Pastena M, Malleo G, Marchegiani G, Butturini G, Violi V, Salvia R, Bassi C. Poor Results of Pancreatoduodenectomy in High-Risk Patients with Endoscopic Stent and Bile Colonization are Associated with E. coli, Diabetes and Advanced Age. J Gastrointest Surg. 2016 Jul;20(7):1359-67. doi: 10.1007/s11605-016-3158-3. Epub 2016 May 11. PMID 27170172
- [Result] Wu JM, Kuo TC, Wu CH, Tien YW. Placement of Nasogastric Tubes in Pancreaticoduodenectomy Patients: Switching from Immediate Intraoperative Removal to Avoiding Unnecessary Perioperative Use. Curr Probl Surg. 2024 Feb;61(2):101439. doi: 10.1016/j.cpsurg.2024.101439. Epub 2024 Jan 10. PMID 38360010
- [Result] Kim HJ, Lee HJ, Cho HJ, Kim HK, Cho AR, Oh N. Nasogastric tube insertion using airway tube exchanger in anesthetized and intubated patients. Korean J Anesthesiol. 2016 Dec;69(6):568-572. doi: 10.4097/kjae.2016.69.6.568. Epub 2016 Sep 28. PMID 27924196
- [Result] Joshi GP, Abdelmalak BB, Weigel WA, Harbell MW, Kuo CI, Soriano SG, Stricker PA, Tipton T, Grant MD, Marbella AM, Agarkar M, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting: Carbohydrate-containing Clear Liquids with or without Protein, Chewing Gum, and Pediatric Fasting Duration-A Modular Update of the 2017 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting. Anesthesiology. 2023 Feb 1;138(2):132-151. doi: 10.1097/ALN.0000000000004381. PMID 36629465
- [Result] Pessaux P, Regimbeau JM, Dondero F, Plasse M, Mantz J, Belghiti J. Randomized clinical trial evaluating the need for routine nasogastric decompression after elective hepatic resection. Br J Surg. 2007 Mar;94(3):297-303. doi: 10.1002/bjs.5728. PMID 17315273
- [Result] Carrere N, Seulin P, Julio CH, Bloom E, Gouzi JL, Pradere B. Is nasogastric or nasojejunal decompression necessary after gastrectomy? A prospective randomized trial. World J Surg. 2007 Jan;31(1):122-7. doi: 10.1007/s00268-006-0430-9. PMID 17186430
- [Result] Rao W, Zhang X, Zhang J, Yan R, Hu Z, Wang Q. The role of nasogastric tube in decompression after elective colon and rectum surgery: a meta-analysis. Int J Colorectal Dis. 2011 Apr;26(4):423-9. doi: 10.1007/s00384-010-1093-4. Epub 2010 Nov 24. PMID 21107848
- [Result] Argov S, Goldstein I, Barzilai A. Is routine use of the nasogastric tube justified in upper abdominal surgery? Am J Surg. 1980 Jun;139(6):849-50. doi: 10.1016/0002-9610(80)90395-5. PMID 7386740
- [Result] Nelson R, Edwards S, Tse B. Prophylactic nasogastric decompression after abdominal surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD004929. doi: 10.1002/14651858.CD004929.pub3. PMID 17636780